CLINICAL TRIAL: NCT03749317
Title: A Double-Masked, Placebo-Controlled, Randomized, Phase II Clinical Trial To Assess The Efficacy Of IVIEW-1201 In The Treatment Of Acute Adenoviral Conjunctivitis
Brief Title: Trial to Evaluate the Efficacy and Safety of IVIEW-1201 in Acute Viral Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IVIEW Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVIEW-1201-01-AIC
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Adenoviral Conjunctivitis
Keywords: IVIEW-1201; Adenoviral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): IVIEW-1201; four times per day (QID) for 7 days
  Interventions: Drug: IVIEW-1201
- Placebo (Placebo Comparator): Placebo; four times per day (QID) for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVIEW-1201 — IVIEW-1201; QID; one drop per eye, four times per day (QID) for 7 days
  Other Names: Treatment Arm
  Arms: Treatment
Drug: Placebo — Placebo drug; QID; one drop per eye, four times per day (QID) for 7 days
  Other Names: Placebo Treatment Arm
  Arms: Placebo

SUMMARY:
A Phase 2, Multi-center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of IVIEW-1201 (1.0% Povidone-Iodine) Gel Forming Ophthalmic Solution Compared to Placebo in the Treatment of Adenoviral Conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
2. Ability to voluntarily provide written, signed, and dated to participate in the study.
3. Subjects of age 15 and over at Visit 1.
4. Have a positive AdenoPlus® test at Visit 1 in at least 1 eye.
5. Have a clinical diagnosis of suspected adenoviral conjunctivitis in at least 1 eye (the same eye as the AdenoPlus positive eye) confirmed by the presence of the following minimal clinical signs and symptoms in that same eye:

   * Reported presence of signs and/or symptoms of adenoviral conjunctivitis for ≤ 3 days prior to Visit 1
   * Bulbar conjunctival injection: a grade of >=1 on 0-4 scale of Bulbar Conjunctival Injection Scale
   * Watery conjunctival discharge: a grade of >=1 (mild) on a 0-3 Watery Conjunctival Discharge Scale
6. Be willing to discontinue contact lens wear for the duration of the study.
7. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria:

Subjects are excluded from the study if any of the following exclusion criteria are met.

1. Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments, per investigator's discretion.
2. Current or relevant history of physical or psychiatric illness, any medical disorder that may make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
3. Have known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
4. Prior enrollment in IVIEW-1201 clinical study.
5. Subjects who are employees, or immediate family members of employees (who are directly related to study conduct), at the investigational site.
6. Have a history of ocular surgical intervention within ≤ 6 months prior to Visit 1 or planned for the period of the study.
7. Have a preplanned overnight hospitalization during the period of the study.
8. Have presence of any intraocular, corneal, or conjunctival ocular inflammation (eg, uveitis, iritis, ulcerative keratitis, chronic blepharoconjunctivitis), other than adenoviral conjunctivitis.
9. Have presence of corneal subepithelial infiltrates at Visit 1
10. Have at enrollment or within ≤30 days of Visit 1, a clinical presentation more consistent with the diagnosis of ocular allergy, toxic conjunctivitis, or non-adenoviral ocular infection (eg, bacterial, fungal, acanthamoebae, other or parasitic).
11. Age under 15.
12. Prisoner.
13. Presence of nasolacrimal duct obstruction at Visit 1 (Day 1).
14. Presence of any significant ophthalmic condition (eg, Retinopathy of Prematurity, congenital cataract, congenital glaucoma) or other congenital disorder with ophthalmic involvement that could affect study variables.
15. Have a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome; presence of corneal epithelial defect or any significant corneal opacity at Visit 1.
16. Presence of significant, active condition in the posterior segment which requires invasive treatment (eg, intravitreal treatment with vascular endothelial growth factor (VEGF) inhibitors or corticosteroids) and may progress during the study participation period.
17. Have used any topical ocular or systemic anti-viral or antibiotics within <= 7 days of enrollment.
18. Have used any topical ocular NSAIDs within <=1 day of enrollment.
19. Have used any topical ophthalmic steroids in the last <=14 days.
20. Have used any systemic corticosteroid agents within <=14 days of Day 1. Stable (initiated ≥30 days prior to enrollment) use of inhaled and nasal corticosteroids is allowed, given no anticipated change in dose for the duration of the study. Topical dermal steroids are allowed except in the peri-ocular area.
21. Have used non-corticosteroid immunosuppressive agents within <=14 days of Day 1, oral or topical or both.
22. Have used any topical ophthalmic products, including tear substitutes, and over-the-counter preparations such as lid scrubs, within 2 hours of Visit 1 and be unable to discontinue all topical ophthalmic products for the duration of the study. Use of hot or cold compresses is also not permitted during the study.
23. Have any significant ocular disease (eg, Sjogren's syndrome) or any uncontrolled systemic disease or debilitating disease (eg, cardiovascular disease, hypertension, sexually transmitted diseases/infections, diabetes or cystic fibrosis), that may affect the study parameters, per Investigator's discretion.
24. Any known history of immunodeficiency disorder or known active conditions predisposing to immunodeficiency, such as human immunodeficiency virus, hepatitis B or C, evidence of active hepatitis A (antihepatitis A virus immunoglobulin M), or organ or bone marrow transplantation.
25. Within 30 days prior to the first dose of investigational product:

    1. Have used an investigational product or device, or
    2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this IVIEW-sponsored study.
26. Pregnant women confirmed with dipstick urine pregnancy testing at Screening and at the final visit.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical resolution by assessment of bulbar conjunctival injection and watery conjunctival discharge | Day 6 +/- 1 Day
  Proportion of subjects achieving clinical resolution (zero for conjunctival injection and discharge)

SECONDARY OUTCOMES:
Viral Eradication | Day 6 +/- 1 Day
  Proportion of subjects with negative cell culture-immunofluorescence assay (CC-IFA)

CONTACTS AND LOCATIONS:
Locations (1):
- Disha Eye Hospital, Kolkata, West Bengal, India